CLINICAL TRIAL: NCT00383292
Title: A Phase 2 Study of LY573636 Administered as an Intravenous Infusion on Day 1 of a 28-Day Cycle as Second-Line Treatment in Patients With Unresectable or Metastatic Melanoma
Brief Title: A Study of Tasisulam in Treating Participants With Malignant Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10409; H8K-MC-JZAF (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-09-29; First posted 2006-10-03 (Estimated); Results first posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — N-((5-bromo-2-thienyl)sulfonyl)-2,4-dichlorobenzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tasisulam (Experimental)
  Interventions: Drug: tasisulam

INTERVENTIONS:
Drug: tasisulam — Tasisulam dose is dependent on participant's height, weight, and gender and is adjusted to target a specific Cmax based on participant laboratory parameters. Tasisulam is administered intravenously every 28 days until disease progression or other criteria for participant discontinuation are met.
  Other Names: LY573636

SUMMARY:
The primary purpose of this study is to determine the objective response rate (complete and partial response) for participants who receive tasisulam after one prior systemic treatment for unresectable or metastatic melanoma.

DETAILED DESCRIPTION:
Participants will receive a 2-hour intravenous infusion of study drug (tasisulam) once every 28 days. Radiological imaging scans will be performed before the first dose of study drug and then after every other treatment. Participants will be assessed for clinical progression at every visit and for response approximately every 56 days (every other cycle).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of malignant melanoma that is unresectable or metastatic (Stage III or IV)
* Have received 1 previous systemic treatment regimen for unresectable or metastatic melanoma. An immunotherapy or antibody-based regimen (including vaccination-based treatments) is not counted as a prior treatment regimen for determining study eligibility, unless it was combined with a chemotherapeutic or targeted anti-cancer drug.
* Have discontinued all previous therapies for cancer, including chemotherapy, radiotherapy, immunotherapy, or other investigational therapy for at least 30 days

Exclusion Criteria:

* Serious pre-existing medical conditions
* Have received two or more previous treatment regimens for unresectable or metastatic melanoma
* Have a second primary cancer (unless disease-free to more than 2 years)
* Active treatment with Warfarin (Coumadin)
* Primary ocular or mucosal melanoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2006-11; Primary Completion 2011-09 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (13):
- United States (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aurora, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lakeland, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pittsburgh, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
- Australia (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coffs Harbour, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wollongong, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Adelaide, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ashford, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nedlands, Western Australia

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Interim analyses of pharmacokinetic (PK) data resulted in adjusted dosing populations to achieve desired concentrations of study drug within the targeted range.
Pre-assignment Details: Study completion was defined as a participant completing 2 cycles of treatment and end of Cycle 2 radiographic assessment of response.
Groups:
- Tasisulam Dose Target 420 μg/mL Cmax: Tasisulam loading dose targeting 420 micrograms/milliliter (μg/mL) maximum concentration (Cmax) at the end of infusion administered as a 2-hour intravenous (IV) infusion on Day 1 of Cycle 1, followed by a chronic dose of 65% of the loading dose on Day 1 of subsequent 21-day cycles (every three weeks).
- Tasisulam Dose Target 360 μg/mL Cmax: Tasisulam loading dose targeting 360 μg/mL Cmax was administered as a 2-hour IV infusion on Day 1 of Cycle 1, followed by a chronic dose of 90% of the loading dose on Day 1 of subsequent 21-day cycles (every three weeks).
- Tasisulam Albumin-Tailored Dose: Tasisulam dose tailored to lean body weight (LBW) and pre-cycle albumin levels (≤420 μg/mL Cmax) was administered as a 2-hour IV infusion on Day 1 of Cycle 1, followed by chronic dosing ranging from 65% to 90% of the loading dose (tailored by the predose serum albumin for that cycle) on Day 1 of subsequent 28-day cycles (every four weeks).
Period: Overall Study
Arm/Group | Tasisulam Dose Target 420 μg/mL Cmax | Tasisulam Dose Target 360 μg/mL Cmax | Tasisulam Albumin-Tailored Dose
Started | 68 | 32 | 30
Received at Least One Dose of Study Drug | 68 | 32 | 30
Completed | 53 | 26 | 22
Not Completed | 15 | 6 | 8
Not completed — Adverse Event | 4 | 1 | 2
Not completed — Death | 3 | 3 | 3
Not completed — Physician Decision | 4 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 2 | 2
Not completed — Other | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study drug.
Groups:
- Tasisulam Dose Target 420 μg/mL Cmax: Tasisulam loading dose targeting 420 μg/mL maximum concentration at the end of infusion (Cmax) administered as a 2-hour intravenous (IV) infusion on Day 1 of Cycle 1, followed by a chronic dose of 65% of the loading dose on Day 1 of subsequent 21-day cycles (every three weeks).
- Total: Total of all reporting groups
Arm/Group | Tasisulam Dose Target 420 μg/mL Cmax | Tasisulam Dose Target 360 μg/mL Cmax | Tasisulam Albumin-Tailored Dose | Total
Number analyzed (Participants) | 68 | 32 | 30 | 130
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.03 (12.68) | 61.60 (15.89) | 61.35 (11.69) | 59.67 (13.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 10 | 9 | 45
  Male | 42 | 22 | 21 | 85
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 67 | 31 | 30 | 128
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39 | 25 | 26 | 90
  Australia | 29 | 7 | 4 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Objective Response Rate (ORR) (Complete Response + Partial Response)
Description: Participants achieved an objective response if they had a best overall response of complete response (CR) or partial response (PR). According to Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1), CR was the disappearance of all non-nodal target lesions, with the short axes of any target lymph node reduced to <10 mm, the disappearance of all non-target lesions, and the normalization of tumor marker levels (if tumor markers were initially above the upper limit of normal); PR was defined as at least a 30% decrease in the sum of the diameters of target lesions (including the short axes of any target lymph node), taking as reference the baseline sum diameter. For each participant who is not known to have died or to have had objective progression of disease as of the data-inclusion cut-off date for a particular analysis, duration of tumor response was to be censored at the date of the participant's last objective tumor assessment prior to that cut-off date.
Time Frame: Baseline to Measured Progressive Disease (up to 60 Months)
Population: All participants who received at least one dose of study drug.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Tasisulam Dose Target 420 μg/mL Cmax | Tasisulam Dose Target 360 μg/mL Cmax | Tasisulam Albumin-Tailored Dose
Number analyzed (Participants) | 68 | 32 | 30
Percentage of Participants | 10 [0 to 20] | 6 [0 to 10] | 7 [0 to 10]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from baseline until measured PD or death from any cause, whichever is first. According to Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1), PD was at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. In addition to the 20% relative increase, the sum must have also demonstrated an absolute increase of at least 5 millimeters (mm). The appearance of 1 or more new lesions and/or unequivocal progression of existing nontarget lesions was also considered progression. Participants without objectively determined PD, who were alive at the end of the follow-up period (or lost to follow-up), were censored on the date of the participant's last complete radiographic tumor assessment; if no baseline or post-baseline radiologic assessment was available, the participant was censored at the date of randomization.
Time Frame: Baseline to Measured Progressive Disease or Death from Any Cause (up to 42 Months)
Population: All participants who received at least one dose of study drug. Participants censored: Tasisulam Target Cmax 420 µg/mL = 10, Tasisulam Target Cmax 360 µg/mL = 8, Albumin-Tailored Dose = 8.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tasisulam Dose Target 420 μg/mL Cmax | Tasisulam Dose Target 360 μg/mL Cmax | Tasisulam Albumin-Tailored Dose
Number analyzed (Participants) | 68 | 32 | 30
Months | 2.8 [1.6 to 4.3] | 2.8 [1.4 to 5.7] | 3.5 [1.9 to 5.7]

3. Secondary Outcome: Percentage of Participants Achieving Complete Response (CR), Partial Response (PR), or Stable Disease (SD) (Clinical Response Rate)
Description: Participants achieved disease control if they had a best overall response of PR, CR or SD. According to RECIST v1.1, CR was the disappearance of all non-nodal target lesions, with the short axes of any target lymph node reduced to <10 mm, the disappearance of all non-target lesions, and the normalization of tumor marker levels (if tumor markers were initially above the upper limit of normal [ULN]); PR was defined as at least a 30% decrease in the sum of the diameters of target lesions (including the short axes of any target lymph node), taking as reference the baseline sum diameter. SD was neither sufficient shrinkage to qualify as PR nor sufficient increase to qualify as PD, taking as reference the smallest sum diameter since treatment started. Clinical Response Rate was calculated as the number of participants who were free from progression (CR+PR+SD) for ≥2 cycles/number of participants who received at least 1 dose of tasisulam.
Time Frame: Baseline to Progressive Disease or Death Due to Any Cause (up to 60 Months)
Population: All participants who received at least one dose of study drug.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Tasisulam Dose Target 420 μg/mL Cmax | Tasisulam Dose Target 360 μg/mL Cmax | Tasisulam Albumin-Tailored Dose
Number analyzed (Participants) | 68 | 32 | 30
Percentage of Participants | 47 [40 to 60] | 47 [30 to 60] | 50 [30 to 70]

4. Secondary Outcome: Pharmacokinetics: Plasma Clearance Rate of Tasisulam
Time Frame: Cycle 1-3, Day 1, 8 and 15: Predose, End of Infusion, and Postinfusion
Population: All participants who received at least one dose of study drug and had evaluable PK data. PK analysis were performed on combined arms for total drug per protocol.
Measure: Geometric Mean (Standard Error); unit: Liters/hour (L/h)
Groups:
- Tasisulam: Tasisulam dose is dependent on participant's height, weight, and gender and is adjusted to target a specific Cmax based on participant laboratory parameters. Participants will receive a 2-hour intravenous infusion of study drug once every 28 days.
Arm/Group | Tasisulam
Number analyzed (Participants) | 127
Liters/hour (L/h) | 0.0275 (3.57)

5. Secondary Outcome: Overall Survival (OS) Time
Description: OS was defined as time from baseline to the date of death from any cause. Participants who were alive at the end of the follow-up period (or lost to follow-up) were censored on the last date the participant was known to be alive.
Time Frame: Baseline to Death from Any Cause (up to 42 Months)
Population: All participants who received at least one dose of study drug. Participants censored: Tasisulam Target Cmax 420 µg/mL = 25, Tasisulam Target Cmax 360 µg/mL = 17, Albumin-Tailored Dose = 17.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tasisulam Dose Target 420 μg/mL Cmax | Tasisulam Dose Target 360 μg/mL Cmax | Tasisulam Albumin-Tailored Dose
Number analyzed (Participants) | 68 | 32 | 30
Months | 10.5 [7.4 to 12.6] | 11.9 [7.1 to NA] — Not estimable based on insufficient number of participants with event data. | 20.1 [11.2 to 22.2]

6. Secondary Outcome: Duration of Overall Objective Response
Description: The duration of response was measured from the date of CR or PR to first date of documented PD or death and was censored at the date of the last assessment for responders who remained alive and did not have documented PD.
Time Frame: Date of Response to Date of Measured PD (up to 1 Year)
Population: All participants who received at least one dose of study drug. Participants censored: Tasisulam Target Cmax 420 µg/mL = 1, Tasisulam Target Cmax 360 µg/mL = 1, Albumin-Tailored Dose = 0.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tasisulam Dose Target 420 μg/mL Cmax | Tasisulam Dose Target 360 μg/mL Cmax | Tasisulam Albumin-Tailored Dose
Number analyzed (Participants) | 68 | 32 | 30
Months | 5.6 [4.3 to 16.1] | 7.2 [NA to NA] — Not estimable based on insufficient number of participants with event data. | 4.1 [3.5 to 4.7]

7. Secondary Outcome: Duration of Stable Disease (SD)
Description: Duration of SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters while on study. SD is measured at the start of the study drug until progressive disease or death due to any cause, whichever is first. Censoring occurred if a participant did not have a complete baseline disease assessment, initiated on another anti-cancer therapy (censored at the date of the last complete objective progression-free disease assessment before initiation of the new therapy), was not known to have died or had objective progression as of the data inclusion cutoff date for analysis.
Time Frame: Baseline to Progressive Disease or Death Due to Any Cause (up to 1 Year)
Population: All participants who received at least one dose of study drug. Participants censored: Tasisulam Target Cmax 420 µg/mL = 6, Tasisulam Target Cmax 360 µg/mL = 5, Albumin-Tailored Dose = 5.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tasisulam Dose Target 420 μg/mL Cmax | Tasisulam Dose Target 360 μg/mL Cmax | Tasisulam Albumin-Tailored Dose
Number analyzed (Participants) | 68 | 32 | 30
Months | 6.9 [4.1 to 8.0] | 6.4 [2.8 to 7.5] | 5.7 [3.8 to 6.6]

8. Secondary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration (Safety: Adverse Events)
Description: Data presented are the number of participants who experienced SAEs considered by the investigator to be related to study drug administration. A summary of SAEs and all other non-serious Adverse Event(s) (AEs), regardless of causality, is located in the Reported Adverse Event module.
Time Frame: Baseline to Study Completion (up to 60 Months)
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Tasisulam Dose Target 420 μg/mL Cmax | Tasisulam Dose Target 360 μg/mL Cmax | Tasisulam Albumin-Tailored Dose
Number analyzed (Participants) | 68 | 32 | 30
Participants | 13 | 6 | 6

9. Secondary Outcome: Health-Related Quality of Life: Functional Assessment of Cancer Therapy-General (FACT-G) Score
Description: FACT-G is a 27-item compilation of general questions divided into 4 primary health-related quality of life (HRQL) domains: Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, and Functional Well-Being. Total scores ranged from 0 to 172; higher scores = better HRQL.
Time Frame: Baseline to Study Completion (up to 60 Months)
Population: All participants who received at least one dose of study drug and had baseline and post baseline FACT-G data. FACT-G analysis was performed on combined arms per protocol.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Tasisulam
Number analyzed (Participants) | 127
Units on a Scale | 80.76 (15.03)

ADVERSE EVENTS:
Arm/Group | Tasisulam Dose Target 420 μg/mL Cmax | Tasisulam Dose Target 360 μg/mL Cmax | Tasisulam Albumin-Tailored Dose
Serious Adverse Events (participants affected / at risk) | 24/68 | 13/32 | 11/30
Other Adverse Events (participants affected / at risk) | 58/68 | 31/32 | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tasisulam Dose Target 420 μg/mL Cmax (N=68) | Tasisulam Dose Target 360 μg/mL Cmax (N=32) | Tasisulam Albumin-Tailored Dose (N=30)
Anaemia (Blood and lymphatic system disorders) | 5 (11) | 2 (3) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 6 (9) | 1 (2) | 4 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (12) | 3 (4) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac ventricular thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Acute abdomen (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 2 (4) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 2 (2) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (4) | 2 (2) | 3 (4)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 2 (9) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral artery thrombosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3)
Hypotension (Vascular disorders) | 3 (3) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Tasisulam Dose Target 420 μg/mL Cmax (N=68) | Tasisulam Dose Target 360 μg/mL Cmax (N=32) | Tasisulam Albumin-Tailored Dose (N=30)
Anaemia (Blood and lymphatic system disorders) | 11 (100) | 4 (21) | 5 (34)
Leukopenia (Blood and lymphatic system disorders) | 5 (46) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (4)
Neutropenia (Blood and lymphatic system disorders) | 9 (36) | 6 (25) | 2 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 13 (62) | 7 (19) | 11 (48)
Tachycardia (Cardiac disorders) | 1 (2) | 0 (0) | 2 (2)
Vision blurred (Eye disorders) | 4 (15) | 1 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 10 (25) | 5 (22) | 7 (25)
Abdominal pain upper (Gastrointestinal disorders) | 2 (8) | 1 (12) | 3 (20)
Constipation (Gastrointestinal disorders) | 14 (45) | 9 (22) | 4 (15)
Diarrhoea (Gastrointestinal disorders) | 20 (62) | 14 (67) | 10 (21)
Dyspepsia (Gastrointestinal disorders) | 8 (59) | 2 (2) | 2 (9)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (50) | 0 (0) | 2 (12)
Nausea (Gastrointestinal disorders) | 17 (74) | 12 (38) | 5 (9)
Stomatitis (Gastrointestinal disorders) | 5 (8) | 6 (43) | 2 (3)
Vomiting (Gastrointestinal disorders) | 7 (9) | 5 (15) | 2 (3)
Asthenia (General disorders) | 2 (5) | 3 (6) | 1 (15)
Axillary pain (General disorders) | 0 (0) | 2 (11) | 0 (0)
Chest pain (General disorders) | 2 (4) | 4 (5) | 2 (4)
Fatigue (General disorders) | 27 (249) | 16 (94) | 11 (71)
Infusion site pain (General disorders) | 8 (14) | 3 (3) | 6 (8)
Injection site pain (General disorders) | 2 (2) | 2 (2) | 1 (1)
Mucosal inflammation (General disorders) | 3 (11) | 0 (0) | 4 (4)
Oedema peripheral (General disorders) | 6 (56) | 2 (13) | 6 (36)
Pain (General disorders) | 3 (19) | 3 (23) | 2 (10)
Pyrexia (General disorders) | 0 (0) | 3 (3) | 4 (6)
Herpes zoster (Infections and infestations) | 3 (12) | 3 (16) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (9) | 0 (0) | 2 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (3) | 2 (12)
Contusion (Injury, poisoning and procedural complications) | 3 (6) | 5 (18) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 2 (5)
Blood alkaline phosphatase increased (Investigations) | 2 (6) | 1 (6) | 2 (20)
Blood creatinine increased (Investigations) | 4 (20) | 2 (11) | 2 (6)
Haemoglobin decreased (Investigations) | 2 (13) | 3 (8) | 1 (6)
Platelet count decreased (Investigations) | 4 (5) | 3 (4) | 1 (3)
Weight decreased (Investigations) | 3 (20) | 3 (15) | 2 (15)
White blood cell count decreased (Investigations) | 1 (2) | 2 (11) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 7 (22) | 5 (20) | 3 (19)
Dehydration (Metabolism and nutrition disorders) | 5 (13) | 2 (6) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 (24) | 0 (0) | 3 (11)
Hypokalaemia (Metabolism and nutrition disorders) | 9 (46) | 6 (32) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (21) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 6 (13) | 0 (0) | 3 (9)
Hypophosphataemia (Metabolism and nutrition disorders) | 4 (15) | 0 (0) | 3 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (100) | 3 (6) | 2 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (45) | 4 (6) | 1 (7)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (14) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (17) | 2 (4) | 1 (14)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (30) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (20) | 4 (11) | 2 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (17) | 2 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (12) | 5 (10) | 2 (8)
Dizziness (Nervous system disorders) | 5 (23) | 5 (8) | 3 (17)
Dysgeusia (Nervous system disorders) | 7 (58) | 7 (46) | 6 (29)
Headache (Nervous system disorders) | 7 (28) | 4 (26) | 1 (7)
Lethargy (Nervous system disorders) | 1 (3) | 2 (2) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 6 (73) | 2 (14) | 1 (24)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (19) | 2 (21) | 3 (34)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (12) | 3 (9)
Confusional state (Psychiatric disorders) | 0 (0) | 3 (7) | 0 (0)
Depression (Psychiatric disorders) | 1 (6) | 0 (0) | 2 (9)
Insomnia (Psychiatric disorders) | 7 (46) | 3 (19) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 2/22 (672) | 1/21 (192)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (25) | 7 (36) | 5 (31)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (63) | 8 (16) | 5 (15)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 (28) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (38) | 3 (39) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (21) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (7) | 2 (3) | 2 (11)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (56) | 3 (16) | 1 (9)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4 (8) | 3 (29) | 3 (9)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (32) | 3 (23) | 1 (2)
Erythema (Skin and subcutaneous tissue disorders) | 2 (8) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (2) | 5 (32)
Rash (Skin and subcutaneous tissue disorders) | 15 (47) | 4 (10) | 6 (49)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (9)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 1 (1)
Phlebitis (Vascular disorders) | 2 (2) | 2 (4) | 2 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days